CLINICAL TRIAL: NCT03436706
Title: Pre-adolescent Stress and Health Study
Status: Withdrawn | Type: Observational
Why Stopped: This study does not qualify as a clinical trial under current NIH guidelines.
Sponsor: Penn State University (Other)
Collaborators: University of Vermont (Other); Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Martha E. Wadsworth, Associate Professor of Psychology, Penn State University
Other Study IDs: STUDY00007585
Record Dates: First submitted 2018-02-10; First posted 2018-02-19 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: The cohort will consist of male and female children ages 11-12 accompanied by a participating parent over the age of 18 years. The family income of participants in this cohort cannot exceed 200% of the federal poverty level established in 2018.
  Interventions: Other: exposure

INTERVENTIONS:
Other: exposure — exposure to chronic stress

SUMMARY:
Aim 1: To characterize allostatic load (AL) biomarkers in a sample of low-income early adolescents (N = 225). How many children living in low-income homes have atypical or out-of-range biomarker levels, on which biomarkers, and in what combinations (Aim 1a)? Do AL biomarker elevations predict physical and mental health problems in early adolescence (Aim 1b)? How much and what type of change in AL biomarkers occurs between ages 11 and 14 (Aim 1c)?

Aim 2: To investigate in the same sample of early adolescents exposed to varying levels of early life stress (ELS), the relative contributions made by ELS, recent (past year), and cumulative (since age 5) stress exposures to initial AL levels at T1 (Aim 2a), and to changes in AL across the two years of the study (Aim 2b).

Aim 3: To explore the extent to which coping resources, including children's coping skills, children's physiologic self-regulation, and parental coping socialization, uniquely and synergistically influence AL levels and accumulations in these early adolescents.

DETAILED DESCRIPTION:
Childhood adversity is associated with premature diseases of aging, most forms of psychopathology, and early mortality, and chronic stress is a critical mechanism of this phenomenon. Biologically informed interventions are sorely needed to break this pernicious cycle, but very little research has examined potentially malleable psychobiological risk and protective processes during childhood that could be leveraged in interventions. Allostatic Load (AL)-the accumulation of biological insults sustained by the body's attempts to maintain homeostasis in the face of chronic stress-is recognized as one such risk process. Most AL research has thus far been conducted with adults, but the emerging research with adolescents suggests that in-depth examination of AL accumulation processes during early adolescence may yield critical insights needed to develop psychobiologically potent interventions. Coping and self-regulation are potential malleable protective processes, but they have not received much attention in AL research to date. This R01 project will therefore examine the accumulation of AL biomarkers in early adolescence, and will test the contributions of stress (early life, cumulative, recent) and of coping resources (coping skills, parent coping socialization, physiologic regulation) to AL accumulation. In addition, we will examine associations between AL and the emergence of premature diseases of aging (e.g., type II diabetes, metabolic syndrome) by mid-adolescence.

Elevated AL biomarkers have been detected in samples of disadvantaged preadolescents (e.g., Evans, 2003; Keller et al., 2012; Rogosch et al. 2011), and are correlated with health problems in this population. Nevertheless, numerous important gaps in our understanding of youth AL processes remain. First, AL is not well characterized in child or adolescent samples. Most existing research involving children focuses only on select aspects of the AL index (such as cortisol), and a comprehensive assessment of the major classes of biomarkers indicated in AL (metabolic, cardiovascular, immunologic, neuroendocrine) in at-risk children is lacking. Second, the absence of clinical benchmarks linking AL to disease in children is a major limiting factor, which coupled with lower base rates of AL-linked diseases in children, calls into question the typical practice of calculating an AL index using adult thresholds (i.e., upper quartile of range). Third, it is unclear to what extent recent and cumulative stressors experienced after the early life period (birth to age 5) contribute to the development of AL over and above early life stress (ELS) in any age group, and many AL studies do not include in-depth assessments of life stress. Fourth, little is known about the extent to which coping resources (youth coping skills, coping socialization) can buffer children from the development and/or worsening of AL over time. This is a critical question as the lead PI's research has shown that coping skills and resources can buffer at-risk children (e.g., in poverty) from common stressors and that coping has effects on primary neuroendocrine mediators of AL such as the HPA (Wadsworth et al., 2016; Bendezu & Wadsworth, 2017).

The present project will build on the unique strengths and capacities of the two PIs and their co-investigator and will include state-of-the-art assessments of stress, coping resources, and AL to fully capture these processes at multiple levels of analysis. Two-hundred 11-12 year old Medicaid-enrolled patients will be recruited by experienced pediatric research nurses at Penn State Hershey Hope Drive Pediatrics. Twenty-five additional 11-12 year old patients whose families are not Medicaid eligible will serve as a middle class comparison group for biomarker benchmarking. This research affiliated pediatrics practice conducts 40,000 patient visits per year and enrolls patients from both rural and urban communities across central PA. Youth will be followed across two years and participate in three annual assessments. Biological samples will include blood draws, overnight urine, and saliva samples taken at each time point. Assessments will further include (a) parent and child Youth Life Stress Interviews to obtain indices of early, recent, and cumulative life stress, and (b) the Trier Social Stress Test to measure adolescent SAM and HPA activation patterns and parent coping socialization. Parent-child parasympathetic co-regulation and reports of psychological symptoms, parenting, parent-child attachment, and coping skills will also be obtained. We will examine levels and correlates of AL biomarkers at T1 as well as predictors of the changes that occur between T1, T2, and T3 (AL accumulation). Study aims are as follows:

Aim 1: To characterize AL biomarkers in a sample of low-income preadolescents (N = 200). How many children living in low-income homes have atypical or out-of-range biomarker levels (as compared to middle class comparison group) (Aim 1a)? Do prior AL biomarker elevations predict physical and mental health problems at age 13-14 (Aim 1b)? How much and what type of change in AL biomarkers occurs between ages 11 and 14 (Aim 1c)?

Aim 2: To investigate in the same sample of preadolescents exposed to varying levels of ELS, the relative contributions made by ELS, recent (past year), and cumulative (since age 5) stress exposures to initial AL levels at T1 (Aim 2a), and to changes in AL across the two years of the study (Aim 2b).

Aim 3: To examine how coping resources, including children's coping skills, children's physiologic self-regulation, parent-child attachment, and parent coping socialization, uniquely and synergistically influence AL levels and accumulations in early adolescence.

ELIGIBILITY:
Inclusion Criteria:

* Child

  * Age: 11-12 years (inclusive) at the time of enrollment
  * Sex: male or female
  * Fluent in written and spoken English

Parent/Guardian

* Age: ≥18 years
* Sex: male or female
* Fluent in written and spoken English
* Families incomes ≤ 200% of the 2018 federal poverty line per table below:

Exclusion Criteria:

Child

* Age: <11 or ≥13 years at the time of enrollment
* Cognitive impairment
* Pregnant (if female)
* Chronic illness (e.g. psychiatric disorder, cancer or heart disease) or any other medical condition that in the opinion of the investigator disqualifies the subject from participation in the research.

Parent/Guardian

* Age: ≥18 years
* Cognitive impairment
* Prisoner

Ages: 132 Months to 156 Months | Sex: All
Age Groups: Child
Study Population: Children living in or near Hershey, Pennsylvania who are living below the federal poverty line. These children and their families are known to experience higher levels of stress the health disparities as a result of living with poverty-related stress.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Allostatic load | 2 years
  represented as individual change across neuroendocrine, autonomic, immunologic, and metabolomic levels among youth from high-risk, rural poor environments

SECONDARY OUTCOMES:
Child health status | 2 years
  Child health status represented by behavioral, psychological, medical, and physical health outcomes affected by allostatic load.

CONTACTS AND LOCATIONS:
Overall Officials: Martha E Wadsworth, PhD, Principal Investigator — Penn State

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Evans GW. A multimethodological analysis of cumulative risk and allostatic load among rural children. Dev Psychol. 2003 Sep;39(5):924-33. doi: 10.1037/0012-1649.39.5.924. PMID 12952404
- [Background] Rogosch FA, Dackis MN, Cicchetti D. Child maltreatment and allostatic load: consequences for physical and mental health in children from low-income families. Dev Psychopathol. 2011 Nov;23(4):1107-24. doi: 10.1017/S0954579411000587. PMID 22018084
- [Background] Abaied JL, Rudolph KD. Mothers as a resource in times of stress: interactive contributions of socialization of coping and stress to youth psychopathology. J Abnorm Child Psychol. 2010 Feb;38(2):273-89. doi: 10.1007/s10802-009-9364-7. PMID 19908139
- [Background] Abaied JL, Rudolph KD. Maternal influences on youth responses to peer stress. Dev Psychol. 2011 Nov;47(6):1776-85. doi: 10.1037/a0025439. Epub 2011 Sep 12. PMID 21910532
- [Background] Grant KE, Compas BE, Thurm AE, McMahon SD, Gipson PY, Campbell AJ, Krochock K, Westerholm RI. Stressors and child and adolescent psychopathology: evidence of moderating and mediating effects. Clin Psychol Rev. 2006 May;26(3):257-83. doi: 10.1016/j.cpr.2005.06.011. Epub 2005 Dec 20. PMID 16364522
- [Background] Wadsworth ME, Rindlaub L, Hurwich-Reiss E, Rienks S, Bianco H, Markman HJ. A longitudinal examination of the Adaptation to Poverty-Related Stress Model: predicting child and adolescent adjustment over time. J Clin Child Adolesc Psychol. 2013;42(5):713-25. doi: 10.1080/15374416.2012.755926. Epub 2013 Jan 16. PMID 23323863
- [Background] Wadsworth ME. Development of Maladaptive Coping: A Functional Adaptation to Chronic, Uncontrollable Stress. Child Dev Perspect. 2015 Jun 1;9(2):96-100. doi: 10.1111/cdep.12112. PMID 26019717
- [Background] Wilkinson RG, Pickett KE. Income inequality and socioeconomic gradients in mortality. Am J Public Health. 2008 Apr;98(4):699-704. doi: 10.2105/AJPH.2007.109637. Epub 2007 Sep 27. PMID 17901426
- [Background] Chen E, Hanson MD, Paterson LQ, Griffin MJ, Walker HA, Miller GE. Socioeconomic status and inflammatory processes in childhood asthma: the role of psychological stress. J Allergy Clin Immunol. 2006 May;117(5):1014-20. doi: 10.1016/j.jaci.2006.01.036. Epub 2006 Mar 9. PMID 16675327
- [Background] Evans, G.W., et al., How poverty gets under the skin: A life course perspective. The Oxford Handbook of Poverty and Child Development, 2012: p. 13-36.
- [Background] Grant, K.E., et al., Protective factors affecting low-income urban African American youth exposed to stress. The Journal of Early Adolescence, 2000. 20(4): p. 388-417.
- [Background] Miech, R.A., et al., Low socioeconomic status and mental disorders: A longitudinal study of selection and causation during young adulthood American Journal of Sociology, 1999. 104(4): p. 1096-1131.
- [Background] Wadsworth ME, Santiago CD. Risk and resiliency processes in ethnically diverse families in poverty. J Fam Psychol. 2008 Jun;22(3):399-410. doi: 10.1037/0893-3200.22.3.399. PMID 18540768
- [Background] McBride Murry, V., et al., Neighborhood poverty and adolescent development. Journal of Research on Adolescence, 2011. 21(1): p. 114-128
- [Background] Wadsworth, M.E., Evans, G.W., Grant, K., Carter, J.S., Duffy, J.S., Poverty and the Development of Psychopathology, in Developmental Psychopathology, D. Cicchetti, Editor 2014.
- [Background] Ackerman BP, Brown ED, Izard CE. The relations between persistent poverty and contextual risk and children's behavior in elementary school. Dev Psychol. 2004 May;40(3):367-77. doi: 10.1037/0012-1649.40.3.367. PMID 15122963
- [Background] Slopen N, Fitzmaurice G, Williams DR, Gilman SE. Poverty, food insecurity, and the behavior for childhood internalizing and externalizing disorders. J Am Acad Child Adolesc Psychiatry. 2010 May;49(5):444-52. doi: 10.1097/00004583-201005000-00005. PMID 20431464
- [Background] Spence SH, Najman JM, Bor W, O'Callaghan MJ, Williams GM. Maternal anxiety and depression, poverty and marital relationship factors during early childhood as predictors of anxiety and depressive symptoms in adolescence. J Child Psychol Psychiatry. 2002 May;43(4):457-69. doi: 10.1111/1469-7610.00037. PMID 12030592
- [Background] Holzer, H.J., et al., The economic costs of childhood poverty in the United States. Journal of Children and Poverty, 2008. 14(1): p. 41-61.
- [Background] Keeshin BR, Cronholm PF, Strawn JR. Physiologic changes associated with violence and abuse exposure: an examination of related medical conditions. Trauma Violence Abuse. 2012 Jan;13(1):41-56. doi: 10.1177/1524838011426152. Epub 2011 Dec 19. PMID 22186168
- [Background] Schreier HM, Schonert-Reichl KA, Chen E. Effect of volunteering on risk factors for cardiovascular disease in adolescents: a randomized controlled trial. JAMA Pediatr. 2013 Apr;167(4):327-32. doi: 10.1001/jamapediatrics.2013.1100. PMID 23440253
- [Background] Gruenewald, T., et al., Socioeconomic gradients in biological markers of disease risk, in Biological Consequences of Socioeconomic Inequalities, The, B. Wolfe, W. Evans, and T.E. Seeman, Editors. 2012, Russell Sage Foundation: New York. p. 63-102.
- [Background] Karlamangla, A.S., T. Gruenewald, and T.E. Seeman, Promise of biomarkers in assessing and predicting health, in The Biological Consequences of Socioeconomic Inequalities, B. Wolfe, W. Evans, and T.E. Seeman, Editors. 2012, Russell Sage Foundation: New York p. 38-62.
- [Background] Chrousos GP. The HPA axis and the stress response. Endocr Res. 2000 Nov;26(4):513-4. doi: 10.3109/07435800009048562. No abstract available. PMID 11196421
- [Background] Goldstein DS. Plasma catecholamines and essential hypertension. An analytical review. Hypertension. 1983 Jan-Feb;5(1):86-99. doi: 10.1161/01.hyp.5.1.86. PMID 6336721
- [Background] Evans GW, Kim P, Ting AH, Tesher HB, Shannis D. Cumulative risk, maternal responsiveness, and allostatic load among young adolescents. Dev Psychol. 2007 Mar;43(2):341-51. doi: 10.1037/0012-1649.43.2.341. PMID 17352543
- [Background] Santiago CD, Wadsworth ME. Family and cultural influences on low-income latino children's adjustment. J Clin Child Adolesc Psychol. 2011;40(2):332-7. doi: 10.1080/15374416.2011.546038. PMID 21391028
- [Background] Wadsworth ME, Achenbach TM. Explaining the link between low socioeconomic status and psychopathology: testing two mechanisms of the social causation hypothesis. J Consult Clin Psychol. 2005 Dec;73(6):1146-53. doi: 10.1037/0022-006X.73.6.1146. PMID 16392987
- [Background] Wadsworth, M.E. and L.E. Berger, Adolescents coping with poverty-related family stress: Prospective predictors of coping and psychological symptoms. Journal of Youth and Adolescence, 2006. 35(1): p. 54-67.
- [Background] Wadsworth, M.E. and B.E. Compas, Coping with family conflict and economic strain: The adolescent perspective. Journal of Research on Adolescence, 2002. 12(2): p. 243-274.
- [Background] Wadsworth, M.E., et al., Adolescent Coping with Poverty-Related Stress. Prevention Researcher, 2008. 15(4): p. 13-16.
- [Background] Wolff BC, Santiago CD, Wadsworth ME. Poverty and involuntary engagement stress responses: examining the link to anxiety and aggression within low-income families. Anxiety Stress Coping. 2009 May;22(3):309-25. doi: 10.1080/10615800802430933. PMID 19253173
- [Background] Attar, B.K., N.G. Guerra, and P.H. Tolan, Neighborhood disadvantage, stressful life events and adjustments in urban elementary-school children. Journal of Clinical Child Psychology, 1994. 23(4): p. 391-400.
- [Background] Bendersky, M. and M. Lewis, Environmental risk, biological risk, and developmental outcome. Developmental Psychology, 1994. 30(4): p. 484.
- [Background] Brooks-Gunn, J., P.K. Klebanov, and F.-R. Liaw, The learning, physical, and emotional environment of the home in the context of poverty: The Infant Health and Development Program. Children and Youth Services Review, 1995. 17(1): p. 251-276.
- [Background] DuBois DL, Felner RD, Meares H, Krier M. Prospective investigation of the effects of socioeconomic disadvantage, life stress, and social support on early adolescent adjustment. J Abnorm Psychol. 1994 Aug;103(3):511-22. doi: 10.1037//0021-843x.103.3.511. PMID 7930051
- [Background] Dubow EF, Tisak J, Causey D, Hryshko A, Reid G. A two-year longitudinal study of stressful life events, social support, and social problem-solving skills: contributions to children's behavioral and academic adjustment. Child Dev. 1991 Jun;62(3):583-99. doi: 10.1111/j.1467-8624.1991.tb01554.x. PMID 1914627
- [Background] McLoyd VC. Socioeconomic disadvantage and child development. Am Psychol. 1998 Feb;53(2):185-204. doi: 10.1037//0003-066x.53.2.185. PMID 9491747
- [Background] Pungello, E.P., et al., Environmental risk factors and children's achievement from middle childhood to early adolescence. Developmental Psychology, 1996. 32(4): p. 755.
- [Background] Evans GW. The environment of childhood poverty. Am Psychol. 2004 Feb-Mar;59(2):77-92. doi: 10.1037/0003-066X.59.2.77. PMID 14992634
- [Background] Evans GW, Li D, Whipple SS. Cumulative risk and child development. Psychol Bull. 2013 Nov;139(6):1342-96. doi: 10.1037/a0031808. Epub 2013 Apr 8. PMID 23566018
- [Background] Obradovic, J., A. Shaffer, and A.S. Masten, Risk in developmental psychopathology: Progress and future directions. The Environment of Human Development: A Handbook of Theory and Measurement, 2012.
- [Background] Sameroff, A., Identifying risk and protective factors for healthy child development. Families Count: Effects on Child and Adolescent Development, 2006: p. 53-76.
- [Background] Evans, G.W., J. Eckenrode, and L.A. Marcynyszyn, Chaos and the macrosetting: The role of poverty and socioeconomic status. 2010.
- [Background] Fiese, B.H., Family routines and rituals2006: Yale University Press.
- [Background] Fiese, B.H. and M.A. Winter, The dynamics of family chaos and its relation to children's socioemotional well-being. 2010.
- [Background] Fuller-Rowell TE, Evans GW, Ong AD. Poverty and health: the mediating role of perceived discrimination. Psychol Sci. 2012 Jul 1;23(7):734-9. doi: 10.1177/0956797612439720. Epub 2012 Jun 14. PMID 22700331
- [Background] Hostinar CE, Lachman ME, Mroczek DK, Seeman TE, Miller GE. Additive contributions of childhood adversity and recent stressors to inflammation at midlife: Findings from the MIDUS study. Dev Psychol. 2015 Nov;51(11):1630-44. doi: 10.1037/dev0000049. Epub 2015 Sep 21. PMID 26389605
- [Background] Piazza JR, Charles ST, Sliwinski MJ, Mogle J, Almeida DM. Affective reactivity to daily stressors and long-term risk of reporting a chronic physical health condition. Ann Behav Med. 2013 Feb;45(1):110-20. doi: 10.1007/s12160-012-9423-0. PMID 23080393
- [Background] Compas BE, Connor-Smith JK, Saltzman H, Thomsen AH, Wadsworth ME. Coping with stress during childhood and adolescence: problems, progress, and potential in theory and research. Psychol Bull. 2001 Jan;127(1):87-127. PMID 11271757
- [Background] Wadsworth, M.E., et al., Parent and adolescent responses to poverty related stress: Tests of mediated and moderated coping models. Journal of Child and Family Studies, 2005. 14(2): p. 283-298.
- [Background] Wadsworth ME, Raviv T, Santiago CD, Etter EM. Testing the adaptation to poverty-related stress model: predicting psychopathology symptoms in families facing economic hardship. J Clin Child Adolesc Psychol. 2011;40(4):646-57. doi: 10.1080/15374416.2011.581622. PMID 21722035
- [Background] Conger, R. and G.H. Elder, Families in troubled times : adapting to change in rural America1994, New York: A. de Gruyter.
- [Background] Santiago, C.D. and M.E. Wadsworth, Coping with family conflict: What's helpful and what's not for low-income adolescents. Journal of Child and Family Studies, 2009. 18(2): p. 192-202.
- [Background] Raviv, T. and M.E. Wadsworth, The efficacy of a pilot prevention program for children and caregivers coping with economic strain. Cognitive Therapy and Research, 2010. 34(3): p. 216-228.
- [Background] Skinner EA, Zimmer-Gembeck MJ. The development of coping. Annu Rev Psychol. 2007;58:119-44. doi: 10.1146/annurev.psych.58.110405.085705. PMID 16903804
- [Background] Abaied, J.L., C. Wagner, and W. Sanders, Parent socialization of coping in emerging adulthood: Moderation by respiratory sinus arrhythmia. Journal of Applied Developmental Psychology, 2014. 35(4): p. 357-369.
- [Background] Kliewer W, Fearnow MD, Miller PA. Coping socialization in middle childhood: tests of maternal and paternal influences. Child Dev. 1996 Oct;67(5):2339-57. PMID 9022245
- [Background] Kliewer W, Parrish KA, Taylor KW, Jackson K, Walker JM, Shivy VA. Socialization of coping with community violence: influences of caregiver coaching, modeling, and family context. Child Dev. 2006 May-Jun;77(3):605-23. doi: 10.1111/j.1467-8624.2006.00893.x. PMID 16686791
- [Background] Miller, P.A., et al., Maternal socialization of children's postdivorce coping: Development of a measurement model. Journal of Applied Developmental Psychology, 1994. 15(3): p. 457-487.
- [Background] Mize J, Pettit GS. Mothers' social coaching, mother-child relationship style, and children's peer competence: is the medium the message? Child Dev. 1997 Apr;68(2):312-32. PMID 9180004
- [Background] Monti JD, Rudolph KD, Abaied JL. Contributions of maternal emotional functioning to socialization of coping. J Soc Pers Relat. 2014 Mar 1;31(2):247-269. doi: 10.1177/0265407513492304. Epub 2013 Jun 25. PMID 26973372
- [Background] Stanger S, Abaied J, Wagner C, Sanders W. Contributions of Observed Parent Socialization of Coping and Skin Conductance Level Reactivity to Childhood Adjustment. Fam Process. 2018 Mar;57(1):181-194. doi: 10.1111/famp.12272. Epub 2016 Dec 18. PMID 27988925
- [Background] Werner NE, Eaton AD, Lyle K, Tseng H, Holst B. Maternal Social Coaching Quality Interrupts the Development of Relational Aggression During Early Childhood. Soc Dev. 2014 Aug 1;23(3):470-486. doi: 10.1111/sode.12048. PMID 25132727
- [Background] Abaied JL, Rudolph KD. Contributions of Maternal Adult Attachment to Socialization of Coping. J Soc Pers Relat. 2010 Aug 1;27(5):637-657. doi: 10.1177/0265407510368966. PMID 21892245
- [Background] Wagner CR, Abaied JL. Relational victimization and proactive versus reactive relational aggression: The moderating effects of respiratory sinus arrhythmia and skin conductance. Aggress Behav. 2015 Nov-Dec;41(6):566-79. doi: 10.1002/ab.21596. Epub 2015 Jul 14. PMID 26174166
- [Background] Abaied, J.L. and C. Emond, Parent Psychological Control and Responses to Interpersonal Stress in Emerging Adulthood Moderating Effects of Behavioral Inhibition and Behavioral Activation. Emerging Adulthood, 2013. 1(4): p. 258-270.
- [Background] Porges SW. The polyvagal perspective. Biol Psychol. 2007 Feb;74(2):116-43. doi: 10.1016/j.biopsycho.2006.06.009. Epub 2006 Oct 16. PMID 17049418
- [Background] Beauchaine T. Vagal tone, development, and Gray's motivational theory: toward an integrated model of autonomic nervous system functioning in psychopathology. Dev Psychopathol. 2001 Spring;13(2):183-214. doi: 10.1017/s0954579401002012. PMID 11393643
- [Background] Alkozei A, Creswell C, Cooper PJ, Allen JJ. Autonomic arousal in childhood anxiety disorders: associations with state anxiety and social anxiety disorder. J Affect Disord. 2015 Apr 1;175:25-33. doi: 10.1016/j.jad.2014.11.056. Epub 2014 Dec 6. PMID 25590763
- [Background] Beauchaine TP, Gatzke-Kopp L, Mead HK. Polyvagal Theory and developmental psychopathology: emotion dysregulation and conduct problems from preschool to adolescence. Biol Psychol. 2007 Feb;74(2):174-84. doi: 10.1016/j.biopsycho.2005.08.008. Epub 2006 Oct 12. PMID 17045726
- [Background] Beauchaine TP, McNulty T. Comorbidities and continuities as ontogenic processes: toward a developmental spectrum model of externalizing psychopathology. Dev Psychopathol. 2013 Nov;25(4 Pt 2):1505-28. doi: 10.1017/S0954579413000746. PMID 24342853
- [Background] Calkins SD, Keane SP. Cardiac vagal regulation across the preschool period: stability, continuity, and implications for childhood adjustment. Dev Psychobiol. 2004 Nov;45(3):101-12. doi: 10.1002/dev.20020. PMID 15505799
- [Background] Gazelle H, Druhen MJ. Anxious solitude and peer exclusion predict social helplessness, upset affect, and vagal regulation in response to behavioral rejection by a friend. Dev Psychol. 2009 Jul;45(4):1077-96. doi: 10.1037/a0016165. PMID 19586181
- [Background] Musser ED, Backs RW, Schmitt CF, Ablow JC, Measelle JR, Nigg JT. Emotion regulation via the autonomic nervous system in children with attention-deficit/hyperactivity disorder (ADHD). J Abnorm Child Psychol. 2011 Aug;39(6):841-52. doi: 10.1007/s10802-011-9499-1. PMID 21394506
- [Background] Posthumus JA, Bocker KB, Raaijmakers MA, Van Engeland H, Matthys W. Heart rate and skin conductance in four-year-old children with aggressive behavior. Biol Psychol. 2009 Oct;82(2):164-8. doi: 10.1016/j.biopsycho.2009.07.003. Epub 2009 Jul 22. PMID 19596046
- [Background] Santucci AK, Silk JS, Shaw DS, Gentzler A, Fox NA, Kovacs M. Vagal tone and temperament as predictors of emotion regulation strategies in young children. Dev Psychobiol. 2008 Apr;50(3):205-16. doi: 10.1002/dev.20283. PMID 18335488
- [Background] Forbes EE, Fox NA, Cohn JF, Galles SF, Kovacs M. Children's affect regulation during a disappointment: psychophysiological responses and relation to parent history of depression. Biol Psychol. 2006 Mar;71(3):264-77. doi: 10.1016/j.biopsycho.2005.05.004. Epub 2005 Aug 22. PMID 16115722
- [Background] Gunnar MR, Frenn K, Wewerka SS, Van Ryzin MJ. Moderate versus severe early life stress: associations with stress reactivity and regulation in 10-12-year-old children. Psychoneuroendocrinology. 2009 Jan;34(1):62-75. doi: 10.1016/j.psyneuen.2008.08.013. Epub 2008 Oct 2. PMID 18835102
- [Background] Lovallo WR. Early life adversity reduces stress reactivity and enhances impulsive behavior: implications for health behaviors. Int J Psychophysiol. 2013 Oct;90(1):8-16. doi: 10.1016/j.ijpsycho.2012.10.006. Epub 2012 Oct 17. PMID 23085387
- [Background] Luecken LJ, Rodriguez AP, Appelhans BM. Cardiovascular stress responses in young adulthood associated with family-of-origin relationship experiences. Psychosom Med. 2005 Jul-Aug;67(4):514-21. doi: 10.1097/01.psy.0000160466.10397.18. PMID 16046362
- [Background] Luecken LJ, Roubinov DS. Hostile behavior links negative childhood family relationships to heart rate reactivity and recovery in young adulthood. Int J Psychophysiol. 2012 May;84(2):172-9. doi: 10.1016/j.ijpsycho.2012.02.003. Epub 2012 Feb 11. PMID 22331058
- [Background] Oosterman M, De Schipper JC, Fisher P, Dozier M, Schuengel C. Autonomic reactivity in relation to attachment and early adversity among foster children. Dev Psychopathol. 2010 Winter;22(1):109-18. doi: 10.1017/S0954579409990290. PMID 20102650
- [Background] Cummings EM, El-Sheikh M, Kouros CD, Keller PS. Children's skin conductance reactivity as a mechanism of risk in the context of parental depressive symptoms. J Child Psychol Psychiatry. 2007 May;48(5):436-45. doi: 10.1111/j.1469-7610.2006.01713.x. PMID 17501724
- [Background] El-Sheikh M, Keiley M, Erath S, Dyer WJ. Marital conflict and growth in children's internalizing symptoms: the role of autonomic nervous system activity. Dev Psychol. 2013 Jan;49(1):92-108. doi: 10.1037/a0027703. Epub 2012 Mar 26. PMID 22448986
- [Background] El-Sheikh M, Keller PS, Erath SA. Marital conflict and risk for child maladjustment over time: skin conductance level reactivity as a vulnerability factor. J Abnorm Child Psychol. 2007 Oct;35(5):715-27. doi: 10.1007/s10802-007-9127-2. Epub 2007 May 15. PMID 17503176
- [Background] Obradovic J, Bush NR, Boyce WT. The interactive effect of marital conflict and stress reactivity on externalizing and internalizing symptoms: the role of laboratory stressors. Dev Psychopathol. 2011 Feb;23(1):101-14. doi: 10.1017/S0954579410000672. PMID 21262042
- [Background] El-Sheikh M, Harger J, Whitson SM. Exposure to interparental conflict and children's adjustment and physical health: the moderating role of vagal tone. Child Dev. 2001 Nov-Dec;72(6):1617-36. doi: 10.1111/1467-8624.00369. PMID 11768136
- [Background] Erath SA, El-Sheikh M, Hinnant JB, Cummings EM. Skin conductance level reactivity moderates the association between harsh parenting and growth in child externalizing behavior. Dev Psychol. 2011 May;47(3):693-706. doi: 10.1037/a0021909. PMID 21142369
- [Background] Erath SA, El-Sheikh M, Mark Cummings E. Harsh parenting and child externalizing behavior: skin conductance level reactivity as a moderator. Child Dev. 2009 Mar-Apr;80(2):578-92. doi: 10.1111/j.1467-8624.2009.01280.x. PMID 19467012
- [Background] Katz LF. Domestic violence and vagal reactivity to peer provocation. Biol Psychol. 2007 Feb;74(2):154-64. doi: 10.1016/j.biopsycho.2005.10.010. Epub 2006 Nov 22. PMID 17118516
- [Background] Katz LF, Gottman JM. Buffering children from marital conflict and dissolution. J Clin Child Psychol. 1997 Jun;26(2):157-71. doi: 10.1207/s15374424jccp2602_4. PMID 9169376
- [Background] Skowron EA, Cipriano-Essel E, Gatzke-Kopp LM, Teti DM, Ammerman RT. Early adversity, RSA, and inhibitory control: evidence of children's neurobiological sensitivity to social context. Dev Psychobiol. 2014 Jul;56(5):964-78. doi: 10.1002/dev.21175. Epub 2013 Oct 19. PMID 24142832
- [Background] El-Sheikh M, Hinnant JB. Marital conflict, respiratory sinus arrhythmia, and allostatic load: interrelations and associations with the development of children's externalizing behavior. Dev Psychopathol. 2011 Aug;23(3):815-29. doi: 10.1017/S0954579411000320. PMID 21756434
- [Background] Slattery MJ, Grieve AJ, Ames ME, Armstrong JM, Essex MJ. Neurocognitive function and state cognitive stress appraisal predict cortisol reactivity to an acute psychosocial stressor in adolescents. Psychoneuroendocrinology. 2013 Aug;38(8):1318-27. doi: 10.1016/j.psyneuen.2012.11.017. Epub 2012 Dec 17. PMID 23253895
- [Background] Gunnar M, Quevedo K. The neurobiology of stress and development. Annu Rev Psychol. 2007;58:145-73. doi: 10.1146/annurev.psych.58.110405.085605. PMID 16903808
- [Background] Wadsworth ME, Bendezu JJ, Loughlin-Presnal J, Ahlkvist JA, Tilghman-Osborne E, Bianco H, Rindlaub L, Hurwich-Reiss E. Unlocking the Black Box: A Multilevel Analysis of Preadolescent Children's Coping. J Clin Child Adolesc Psychol. 2018 Jul-Aug;47(4):527-541. doi: 10.1080/15374416.2016.1141356. Epub 2016 Mar 30. PMID 27029784
- [Background] Romeo RD, McEwen BS. Stress and the adolescent brain. Ann N Y Acad Sci. 2006 Dec;1094:202-14. doi: 10.1196/annals.1376.022. PMID 17347352
- [Background] Connor-Smith JK, Compas BE, Wadsworth ME, Thomsen AH, Saltzman H. Responses to stress in adolescence: measurement of coping and involuntary stress responses. J Consult Clin Psychol. 2000 Dec;68(6):976-92. PMID 11142550
- [Background] Boxer P, Sloan-Power E, Schappell IM. Coping with stress, coping with violence: Links to mental health outcomes among at-risk youth. J Psychopathol Behav Assess. 2012 Sep 1;34(3):405-414. doi: 10.1007/s10862-012-9285-6. Epub 2012 Apr 19. PMID 23002323
- [Background] Santiago, C.D., M.E. Wadsworth, and J. Stump, Socioeconomic status, neighborhood disadvantage, and poverty-related stress: Prospective effects on psychological syndromes among diverse low-income families. Journal of Economic Psychology, 2011. 32(2): p. 218-230.
- [Background] Wadsworth, M.E., Preadolescents' recovery from acute stress: Timing, context, and correlates of SNS-HPA co-activation. Psychoneuroendocrinology, 2015. 61: p. 38-39.
- [Background] Stanger S, Abaied J, Wagner C. Predicting Heavy Alcohol Use in College Students: Interactions Among Socialization of Coping, Alcohol Use Onset, and Physiological Reactivity. J Stud Alcohol Drugs. 2016 May;77(3):483-94. doi: 10.15288/jsad.2016.77.483. PMID 27172581
- [Background] Wagner CR, Abaied JL. Skin Conductance Level Reactivity Moderates the Association Between Parental Psychological Control and Relational Aggression in Emerging Adulthood. J Youth Adolesc. 2016 Apr;45(4):687-700. doi: 10.1007/s10964-016-0422-5. Epub 2016 Jan 13. PMID 26762376
- [Background] Losoya, S., N. Eisenberg, and R.A. Fabes, Developmental issues in the study of coping. International Journal of Behavioral Development, 1998. 22(2): p. 287-313.
- [Background] Seiffge-Krenke I, Aunola K, Nurmi JE. Changes in stress perception and coping during adolescence: the role of situational and personal factors. Child Dev. 2009 Jan-Feb;80(1):259-79. doi: 10.1111/j.1467-8624.2008.01258.x. PMID 19236405
- [Background] Windle M, Spear LP, Fuligni AJ, Angold A, Brown JD, Pine D, Smith GT, Giedd J, Dahl RE. Transitions into underage and problem drinking: developmental processes and mechanisms between 10 and 15 years of age. Pediatrics. 2008 Apr;121 Suppl 4(Suppl 4):S273-89. doi: 10.1542/peds.2007-2243C. PMID 18381494
- [Background] Hostinar CE, Sullivan RM, Gunnar MR. Psychobiological mechanisms underlying the social buffering of the hypothalamic-pituitary-adrenocortical axis: a review of animal models and human studies across development. Psychol Bull. 2014 Jan;140(1):256-82. doi: 10.1037/a0032671. Epub 2013 Apr 22. PMID 23607429
- [Background] Stroud LR, Papandonatos GD, Williamson DE, Dahl RE. Sex differences in cortisol response to corticotropin releasing hormone challenge over puberty: Pittsburgh Pediatric Neurobehavioral Studies. Psychoneuroendocrinology. 2011 Sep;36(8):1226-38. doi: 10.1016/j.psyneuen.2011.02.017. Epub 2011 Apr 13. PMID 21489699
- [Background] Hankin BL, Abramson LY, Moffitt TE, Silva PA, McGee R, Angell KE. Development of depression from preadolescence to young adulthood: emerging gender differences in a 10-year longitudinal study. J Abnorm Psychol. 1998 Feb;107(1):128-40. doi: 10.1037//0021-843x.107.1.128. PMID 9505045
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Rudolph KD, Flynn M. Childhood adversity and youth depression: influence of gender and pubertal status. Dev Psychopathol. 2007 Spring;19(2):497-521. doi: 10.1017/S0954579407070241. PMID 17459181
- [Background] Brown GW, Harris T. Social origins of depression: a reply. Psychol Med. 1978 Nov;8(4):577-88. doi: 10.1017/s0033291700018791. PMID 724871
- [Background] Abaied, J.L. and K.D. Rudolph, Family relationships, emotional processes, and adolescent depression. The Oxford Handbook of Depression and Comorbidity, 2014: p. 460-475.
- [Background] Flynn M, Rudolph KD. Stress generation and adolescent depression: contribution of interpersonal stress responses. J Abnorm Child Psychol. 2011 Nov;39(8):1187-98. doi: 10.1007/s10802-011-9527-1. PMID 21647600
- [Background] Flynn M, Rudolph KD. The trade-offs of emotional reactivity for youths' social information processing in the context of maternal depression. Front Integr Neurosci. 2012 Jul 13;6:43. doi: 10.3389/fnint.2012.00043. eCollection 2012. PMID 22876221
- [Background] Rudolph KD, Troop-Gordon W, Flynn M. Relational victimization predicts children's social-cognitive and self-regulatory responses in a challenging peer context. Dev Psychol. 2009 Sep;45(5):1444-54. doi: 10.1037/a0014858. PMID 19702404
- [Background] Murray-Close D. Autonomic reactivity and romantic relational aggression among female emerging adults: moderating roles of social and cognitive risk. Int J Psychophysiol. 2011 Apr;80(1):28-35. doi: 10.1016/j.ijpsycho.2011.01.007. Epub 2011 Jan 18. PMID 21251934